CLINICAL TRIAL: NCT05681299
Title: Effects of Administration of Growth Hormone, Without and With Liraglutide, on AgRP, Energy and Glucose Metabolism in Healthy and GH Deficient Humans
Brief Title: Effects of GH and Lirglutide on AgRP
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Pamela U. Freda, Professor of Medicine at CUIMC, Columbia University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: AAAU4280
Record Dates: First submitted 2022-12-27; First posted 2023-01-12 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Healthy; Growth Hormone Deficiency
Keywords: growth hormone; liraglutide; AgRP
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Growth Hormone; Liraglutide

STUDY DESIGN:
Intervention Model Description: Participant blind
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Growth hormone (Active Comparator): GH will be administered as one nightly subcutaneous self-injection at 11pm at a dose of 0.03 mg/kg/day in healthy and 0.5 mg in male and 0.6 mg in female GHD subjects. Injections will be performed from the night of day 0 to the night of day 20.
  Interventions: Drug: growth hormone
- Liraglutide (Active Comparator): Liraglutide will be administered by subcutaneous injection taken by subjects beginning at a dose at 0.6 mg nightly from 9-11 pm and escalated in 0.6 mg increments weekly as tolerated to a final dose of 1.8 mg nightly. Injections will be performed from the night of day 0 to the night of day 20.
  Interventions: Drug: liraglutide
- Growth hormone and liraglutide (Active Comparator): GH will be administered as one nightly subcutaneous self-injection at 11pm at a dose of 0.03 mg/kg/day in healthy and 0.5 mg in male and 0.6 mg in female GHD subjects. Liraglutide will be administered by subcutaneous injection taken by subjects beginning at a dose at 0.6 mg nightly from 9-11 pm and escalated in 0.6 mg increments weekly as tolerated to a final dose of 1.8 mg nightly.
  Injections will be performed from the night of day 0 to the night of day 20.
  Interventions: Drug: growth hormone and lirglutide
- Placebo (Placebo Comparator): Placebo will be administered as one nightly subcutaneous self-injection at 9-11pm from the night of day 0 to the night of day 20.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: growth hormone and lirglutide — GH will be administered as one nightly subcutaneous self-injection at 11pm at a dose of 0.03 mg/kg/day in healthy and 0.5 mg in male and 0.6 mg in female GHD subjects and liraglutide will be administered by subcutaneous injection taken by subjects beginning at a dose at 0.6 mg nightly from 9-11 pm and escalated in 0.6 mg increments weekly as tolerated to a final dose of 1.8 mg nightly.
  Arms: Growth hormone and liraglutide
Drug: growth hormone — GH will be administered as one nightly subcutaneous self-injection at 11pm at a dose of 0.03 mg/kg/day in healthy and 0.5 mg in male and 0.6 mg in female GHD subjects.
  Arms: Growth hormone
Drug: liraglutide — Liraglutide will be administered by subcutaneous injection taken by subjects beginning at a dose at 0.6 mg nightly from 9-11 pm and escalated in 0.6 mg increments weekly as tolerated to a final dose of 1.8 mg nightly.
  Arms: Liraglutide
Drug: Placebo — Placebo will be taken by nightly subcutaneous injection at 9-11 pm.
  Arms: Placebo

SUMMARY:
This is a randomized, placebo-controlled, cross-over study with 4 arms. Healthy and GH deficient adults ages 18-45 years will be studied. Arms will consist of 21-day treatment periods and be separated by 8-week washout periods. Subjects will receive, in random order: i) GH alone, ii) GH with liraglutide, iii) liraglutide alone and iv) placebo. Each phase of the study will consist of a 7-day baseline period including 2 days of testing and 21 days on therapy with visits on days 2, 7, 14 and 21. Testing before, during and at the completion of each arm will include blood sampling and assessments of insulin resistance, energy expenditure and body composition.

DETAILED DESCRIPTION:
Rationale: GH and IGF-1 are vital to growth and metabolism across the human lifespan. In disorders of GH/IGF-1 excess and deficiency and the many other disease processes that perturb these hormones, significant growth and metabolic abnormalities can develop. GH is known to act on peripheral tissues, but recent data suggest that central effects of GH on the orexigenic hypothalamic neuropeptide AgRP (agouti-related peptide) is another important mechanism by which GH exerts its nutritional and metabolic effects. AgRP neurons express GH receptors and, in mice, GH was shown to activate AgRP neurons to produce orexigenic responses. GH may signal nutrient status via AgRP neurons. Our data in patients with acromegaly suggests that GH increases AgRP, but whether GH stimulates AgRP has not been tested. Therefore, this project directly tests that GH administration stimulates AgRP in humans. To further investigate the GH-AgRP axis, this project also tests the effect of the GLP-1R agonist liraglutide on plasma AgRP levels and explores the potential link of GH-stimulated changes in AgRP to GH-induced insulin resistance.

Study population and Design: The study population will include 40 healthy and 24 GH deficient adults. Each group will be half female and all will be between the ages of 18-45 years. The study is a randomized, participant-blind, placebo-controlled cross-over study of four arms: GH, GH+liraglutide, liraglutide and placebo, that are each 3 weeks and separated by an 8-week washout period. Each phase of the study will consist of a 7-day baseline period including 2 days of testing and 21 days on therapy with visits on days 2, 7, 14 and 21. We will apply a Williams cross-over design and randomization procedure(1) to ensure balance within and across groups. Subjects will take nightly subcutaneous injections of study medications or placebo during each arm. Participants will undergo anthropometric measurements and fasting blood sampling at every visit, an oral glucose tolerance test before and at the day 14 visit and assessments of body composition by quantitative magnetic resonance (QMR), energy expenditure and insulin sensitivity before and at the end of each arm. They will complete food and activity recording daily throughout the study except on study visit days.

ELIGIBILITY:
Inclusion Criteria:

HEALTHY SUBJECTS

1. 40 healthy subjects, 20 male, 20 female, ages 18-45 yr.: (i) 20 (10 male, 10 female) who are overweight/Class 1 Obese (BMI 25-34.9) with abdominal fat accumulation (central adiposity) defined by waist circumference (WC) ≥ 102 cm in men, ≥ 88 cm in women, except in East/South Asians for whom the criteria will be WC ≥ 90 men and ≥ 80 women; (ii) 20 (10 male,10 female) who are lean (BMI 19-24.9) and not meeting these WC criteria.
2. No medical conditions except being overweight/obese in half of subjects
3. No prescription medication or other drug use
4. On screening testing: BP<140/<90 mmHg, HbA1c<5.7%, FPG<100 mg/dL, normal IGF-1 and TSH levels.
5. Premenopausal women: use of nonhormonal method of contraception
6. Current non-smoker

GH DEFICIENT SUBJECTS

1. 24 patients with isolated GH deficiency:12 males, 12 females.
2. Ages 18-45 years
3. Diagnosis of isolated GH deficiency based on accepted, BMI-appropriate GH stimulation test cut offs within 12 months of enrollment
4. No prior GH therapy within 12 months of study enrollment
5. Normal thyroid, adrenal and gonadal function documented by accepted stimulation test and clinical criteria
6. Premenopausal women: use of nonhormonal method of contraception

Exclusion Criteria:

HEALTHY SUBJECTS

1. History of malignancy, diabetes, thyroid cancer or pancreatitis
2. Recent dieting, weight change >5%, pregnancy or lactation or heavy exercise
3. Use of glucocorticoids, hormonal supplements or medications that could affect GH or IGF-1 or for weight loss within 6 months of enrollment

GH DEFICIENT SUBJECTS

1. DM requiring medication
2. HbA1C > 7.5
3. Malignancy, pancreatitis or thyroid cancer history.
4. Deficiency of other pituitary hormones, liver or renal disease
5. Use of glucocorticoids, hormonal supplements or medications that could affect GH or IGF-1 or for weight loss within 6 months of enrollment

5. Recent dieting, weight change > 5%, pregnancy, lactation or heavy exercise 6. Current smoking

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
AgRP change in GH vs. placebo arms | Baseline to weeks 1, 2, 3 of each study arm.
  Difference in percent change in morning fasting level of AgRP (agouti-related peptide) in plasma in GH vs. placebo arms.
AgRP change in GH vs. GH + liraglutide arms | Baseline to weeks 1, 2, 3 of each study arm.
  Difference in percent change in morning fasting level of AgRP in plasma in GH vs. GH+liraglutide arms.

SECONDARY OUTCOMES:
AgRP change in GH arm | Baseline to week 1,2, 3 of study arm.
  Percent change in plasma AgRP level with GH therapy
AgRP change in liraglutide vs. placebo arms | Baseline to weeks 1,2, 3 of each study arm
  Difference in percent change in morning fasting level of AgRP in placebo vs. liraglutide arms.

CONTACTS AND LOCATIONS:
Locations (1):
- Neuroendocrine Unit and Pituitary Center, Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No